CLINICAL TRIAL: NCT05695781
Title: A Multi-Center, Randomized, Double Masked, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of BRM421 Ophthalmic Solution in Subjects With Dry Eye Using a Controlled Adverse Environment (CAE®) Model
Brief Title: Assessment of the Safety and Efficacy of BRM421 Ophthalmic Solutions in Dry Eye Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BRIM Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM421-22-C001-PR
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double Masking
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRM421 Ophthalmic Solution (Active Comparator)
  Interventions: Drug: BRM421 Ophthalmic Solution
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BRM421 Ophthalmic Solution — A topical drop of BRM421 ophthalmic solution.
  Arms: BRM421 Ophthalmic Solution
Drug: Vehicle — A topical drop of vehicle (minus active) ophthalmic solution.
  Arms: Vehicle

SUMMARY:
The objective of this study is to compare the safety and efficacy of BRM421 OS to vehicle for the treatment of the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye prior to enrollment;
* Have a history of use or desire to use eye drops;

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Ocular Sign: Change From Baseline in Total Corneal Fluorescein Staining Score | 1-2 weeks
  0-12 Ora scale, higher scores mean a worse outcome.
Ocular Symptom: Change From Baseline in Visual Analog Scale (VAS) | 1-2 weeks
  0-100 Visual Analog Scale, higher scores mean a worse discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Warwick, Rhode Island, United States